CLINICAL TRIAL: NCT00460447
Title: Gentuzumab Ozogamicin Berfore Allogeneic Stem Cell Transplantation in Patients With Relapsed CD33+ Acute Myeloid Leukemia
Brief Title: Gemtuzumab Ozogamicin Before Allogeneic Stem Cell Transplantation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Carl Gustav Carus (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EK 92062003
Record Dates: First submitted 2007-04-12; First posted 2007-04-16 (Estimated); Last update posted 2007-04-16 (Estimated); Status verified 2007-04

CONDITIONS: Acute Myeloid Leukemia; Allogeneic Transplantation
Keywords: anti-CD33; Immunotoxin; Acute myeloid leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Gemtuzumab Ozogamicin

SUMMARY:
Study Design:

prospective phase II trial with 30 patients in 1 site

Treatment Scheme:

Option 1: Patient < 60 years of age with relapse after chemotherapy or > 12 months after hematopoetic stem cell transplantation Mylotarg 6 mg/ m² day -21 Mylotarg 3 mg/ m² day -14 Fludarabin 30 mg/ m² day -6 to -3 TBI 2x2 Gy day -3 to -2 (total dose 8 Gy) Tacrolimus (level adapted) from day -3 on Mycophenolat 2 x 1000 mg p.o. from day 0 to day 40 PBSC day 0

Option 2: Patient > 60 years of age or younger patients < 12 Months after hematopoetic stem cell transplantation Mylotarg 6 mg/ m² day -21 Mylotarg 3 mg/ m² day -14 Fludarabin 30 mg/ m² day -3 to -1 TBI 1x2 Gy day 0 (total dose 2 Gy) Tacrolimus (level adapted) from day -3 on Mycophenolat 2 x 1000 mg p.o. from day 0 to 40 PBSC day 0

DETAILED DESCRIPTION:
Scientific/Medical Rationale (Objective):

Primary:

documentation of the extramedullary toxicity of the standard therapy

Secondary:

Induction of a persistent remission by the combination of Mylotarg and dose reduced conditioning followed by allogenic hematopoetic stem cell transplantation in patients with relapsed acute myelotic leukemia

Study Design:

prospective phase II trial with 30 patients in 1 site

Treatment Scheme:

Option 1: Patient < 60 years of age with relapse after chemotherapy or > 12 months after hematopoetic stem cell transplantation Mylotarg 6 mg/ m² day -21 Mylotarg 3 mg/ m² day -14 Fludarabin 30 mg/ m² day -6 to -3 TBI 2x2 Gy day -3 to -2 (total dose 8 Gy) Tacrolimus (level adapted) from day -3 on Mycophenolat 2 x 1000 mg p.o. from day 0 to day 40 PBSC day 0

Option 2: Patient > 60 years of age or younger patients < 12 Months after hematopoetic stem cell transplantation Mylotarg 6 mg/ m² day -21 Mylotarg 3 mg/ m² day -14 Fludarabin 30 mg/ m² day -3 to -1 TBI 1x2 Gy day 0 (total dose 2 Gy) Tacrolimus (level adapted) from day -3 on Mycophenolat 2 x 1000 mg p.o. from day 0 to 40 PBSC day 0

Patient Population to be Included:

30 patients

Primary and Secondary Efficacy Endpoints:

See point: Scientific/Medical Rationale

Inclusion Criteria /Exclusion Criteria:

* patients with acute myelotic leukemia and expression of CD33 on > 5% of blasts in bone marrow
* relapse after chemotherapy
* relapse after autologous or allogenic hematopoetic stem cell transplantation
* pts. in  2nd remission after chemotherapy and ineligible for a conventional allogeneic transplantation
* age: 18-70 years
* informed consent of the patient
* ASAT/ ALAT < 3fold of upper standard
* Bilirubin < 2fold of upper standard
* ejection fraction > 40% in echocardiography
* potential donor in accordance with the following priorities:
* 1st HLA-identical related donor (HLA *A, *B, *C and *DR)
* 2nd HLA-identical non-related donor with the maximum of 1 allelmismatch (DNA typing A, B, C, DRB1, DQB1)

Study Procedures:

See point . Study Design

Safety Endpoints/ Statistical Considerations:

Thirty patients will be treated, which will yield a 95% confidence interval for non-relapse mortality with a precision of +/- 14%. Data will be evaluated after groups of 10 and 20 patients. If results at those times suggest with greater than 80% confidence that the true rate of day 100 non-relapse mortality exceeds 20%, then the trial will be stopped. Operationally, this will occur if 4 out of 10 or 7 out of 20 patients have non-relapse deaths. Should the requisite number of deaths be reached before the 10 or 20 patient benchmarks, then the trial will be stopped at that time.

A dose reduction of mylotarg from 9 to 6 mg/m2 will be performed if the likelihood of grade 4 liver-toxicity as defined by bilirubine, AST and symptoms of sinusoidal obstruction syndrome is > 20%. This will be the case if 4 out of the first ten patients experience grade 4 liver toxicity. The second dose of mylotarg will then be omitted in the next ten patients. If the rate of liver-toxicity in the next 10 patients remains unchanged, the study will be stopped.

The stopping rules will be discussed and enforced by the protocol committee and transmitted to each local IRB asap.

The following safety endpoints will be documented:

1. Incidence of neurological toxicity
2. Incidence of liver toxicity
3. Incidence of acute gastrointestinal toxicity
4. Incidence and severity of mucositis
5. Incidence of pulmonary toxicity
6. Incidence of systemic infections
7. Duration of neutropenia Severe adverse events (SAE) will have to be reported to the principal investigator within 24 hours after occurrence. It will be his responsibility to inform the IRB and the sponsor or the trial, if adequate.

SAE compromise: death before relapse of leukemia, illness with life-threatening character, severe illness requiring hospitalization, illness leading to prolonged disabilities, second cancer developing after treatment.

SAE will have to be reported on special forms contained in the CRF

ELIGIBILITY:
Inclusion Criteria:

* - patients with acute myelotic leukemia and expression of CD33 on > 5% of blasts in bone marrow
* relapse after chemotherapy
* relapse after autologous or allogenic hematopoetic stem cell transplantation
* pts. in 2nd remission after chemotherapy and ineligible for a conventional allogeneic transplantation
* age: 18-70 years
* informed consent of the patient
* ASAT/ ALAT < 3fold of upper standard
* Bilirubin < 2fold of upper standard
* ejection fraction > 40% in echocardiography
* potential donor in accordance with the following priorities:
* 1st HLA-identical related donor (HLA *A, *B, *C and *DR)
* 2nd HLA-identical non-related donor with the maximum of 1 allelmismatch (DNA typing A, B, C, DRB1, DQB1)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-10

PRIMARY OUTCOMES:
Documentation of the extramedullary toxicity of the standard therapy

SECONDARY OUTCOMES:
Induction of a persistent remission by the combination of Mylotarg and dose reduced conditioning followed by allogenic hematopoetic stem cell transplantation in patients with relapsed acute myelotic leukemia

CONTACTS AND LOCATIONS:
Overall Officials: Martin Bornhäuser, MD, Principal Investigator — Medical Clinic, University Hospital Dresden
Locations (1):
- Medizinische Klinik und Poliklinik I, Dresden, Germany